CLINICAL TRIAL: NCT01919398
Title: A Phase 1 Study of LY2940680 in Japanese Patients With Advanced Solid Tumors
Brief Title: A Study of LY2940680 in Japanese Participants With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14895 TRANSFERRED; I4J-MC-HHBH (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-08-05; First posted 2013-08-09 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — LY2940680

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2940680 (Experimental): Cohort 1: 100 mg LY2940680 administered orally daily in 28-day cycles. Cohort 2: 200 mg LY2940680 administered orally daily in 28-day cycles. Cohort 3: 400 mg LY2940680 administered orally daily in 28-day cycles.
  Treatment with LY2940680 continued until disease progression, unacceptable toxicity, or other discontinuation criteria were met.
  Interventions: Drug: LY2940680

INTERVENTIONS:
Drug: LY2940680 — Administered orally

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of LY2940680 up to the global recommended dose in Japanese participants with advanced solid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of solid tumor that is advanced and/or metastatic. The participant must be, in the judgment of the investigator, an appropriate candidate for the experimental therapy after available standard therapies have failed to provide clinical benefit for their disease
* Have the presence of measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors Guideline Version 1.1
* Have adequate organ function
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy for at least 3 weeks (6 weeks for mitomycin-C or nitrosoureas, 2 weeks for palliative radiation therapy for bone metastasis) prior to study enrollment, and have recovered from the acute effects of any such therapy
* Males must agree to use medically approved barrier contraceptive precautions during the study and for 6 months following the last dose of study drug
* Females with child bearing potential must agree to use medically approved contraceptive precautions during the study and for 6 months following the last dose of study drug; have had a negative serum pregnancy test ≤7 days before the first dose of study drug
* A breastfeeding woman must not be breastfeeding. If a female who stops breastfeeding enters the study, the female must stop breastfeeding from the day of the first study drug administration until at least 6 months after the last administration
* Have an estimated life expectancy, in the judgment of the investigator, which will permit the participant to complete 2 cycles of treatment
* Are able to swallow tablets

Exclusion Criteria:

* Have received treatment within 21 days of the study enrollment with any agent that has not received regulatory approval for any indication
* Have symptomatic central nervous system (CNS) malignancy or metastasis. Participants with treated brain metastases are eligible if they are clinically stable with regard to neurologic function and off steroids after cranial irradiation ending at least 14 days prior to enrollment, or after surgical resection performed at least 28 days prior to enrollment
* Have known current hematologic malignancies or acute or chronic leukemia
* Have a known active fungal, bacterial, and/or known viral infection including human immunodeficiency (HIV) or viral (A, B, or C) hepatitis, potentially affecting the conduct of this study
* Have a second primary malignancy that in the judgment of the investigator and sponsor may affect the interpretation of results
* Have QTc interval of >470 milliseconds (msec) on screening electrocardiogram (ECG)
* Have serious preexisting medical conditions or serious concomitant systemic disorders that, in the opinion of the investigator, would preclude participation in this study
* Have received any medication that is a strong inhibitor of cytochrome P4503A4 (CYP3A4) within 7 days prior to receiving study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 1-858-255-5959 Mon-Fri from 9 AM to 5 PM Pacific Time (PST), Study Director — Hoffmann-La Roche
Locations (2):
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-858-255-5959 Mon - Fri from 9 AM to 5 PM Pacific Time (PST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-858-255-5959 Mon - Fri from 9 AM to 5 PM Pacific Time (PST), or speak with your personal physician., Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study completers were participants who were Dose-Limiting Toxicities (DLT) evaluable and discontinued the treatment due to any reason.
Groups:
- Cohort 1: 100 mg LY2940680: Cohort 1: 100 mg LY2940680 administered orally once daily in 28-day cycles.
  Treatment with LY2940680 continued until disease progression, unacceptable toxicity, or other discontinuation criteria were met.
- Cohort 2: 200 mg LY2940680: Cohort 2: 200 mg LY2940680 administered orally daily in 28-day cycles.
  Treatment with LY2940680 continued until disease progression, unacceptable toxicity, or other discontinuation criteria were met.
- Cohort 3: 400 mg LY2940680: Cohort 3: 400 mg LY2940680 administered orally once daily in 28-day cycles.
  Treatment with LY2940680 continued until disease progression, unacceptable toxicity, or other discontinuation criteria were met.
Period: Overall Study
Arm/Group | Cohort 1: 100 mg LY2940680 | Cohort 2: 200 mg LY2940680 | Cohort 3: 400 mg LY2940680
Started | 3 | 3 | 13
Received at Least One Dose of Study Drug | 3 | 3 | 13
Completed | 3 | 3 | 9
Not Completed | 0 | 0 | 4
Not completed — Progressive Disease | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 100 mg LY2940680 | Cohort 2: 200 mg LY2940680 | Cohort 3: 400 mg LY2940680 | Total
Number analyzed (Participants) | 3 | 3 | 13 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (7.02) | 72.0 (4.36) | 60.7 (11.93) | 62.9 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 1 | 2 | 13 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 13 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3 | 3 | 13 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With LY2940680 Dose-Limiting Toxicities (DLT)
Description: DLT was defined as an AE during Cycle 1 that is possibly related to the study drug and meets any one of the following criteria based on NCI CTCAE,version 4.0): Grade(Gr) 3 nonhematological toxicity(tox) with exceptions for made for nausea(ns),vomiting(vm),constipation(cp),diarrhea(dr),fatigue(ft),anorexia(an),alopecia or electrolyte-abnormality(eab) that is manageable with appropriate care.If >Gr 3 ns,vm,cp,dr,ft,an,or eab persists for>2 days with maximal supportive intervention,the event was declared a DLT.Transient(≤5 days) Gr 3 liver enzyme elevations,without evidence of other hepatic injury.Gr 3 thrombocytopenia(throm) requiring platelet transfusion or Gr 4 throm.Gr 4 neutropenia of >5 days duration.Febrile neutropenia(ANC<1,000/mm3 with a single temperature(temp) of >38.3 degrees C or a sustained temp of ≥38 degrees C for more than one hour).Tox requiring dose omissions of >5 days or significant & deemed by the primary investigator(PI) & sponsor(sp) to be dose limiting .
Time Frame: Cycle 1 (28 Days)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 100 mg LY2940680 | Cohort 2: 200 mg LY2940680 | Cohort 3: 400 mg LY2940680
Number analyzed (Participants) | 3 | 3 | 13
Participants | 0 | 0 | 3

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2940680 and a Major Metabolite of LY2940680 (LSN3185556)
Description: Maximum Concentration (Cmax) of LY2940680 and a Major Metabolite of LY2940680 (LSN3185556).
Time Frame: Cycle1 Day1: Predose, 0.5,1,2,4, 6, 8, 10-12 hours; Cycle 1 Day15: Predose, 0.5,1,2,4, 6, 8, 10-12 hours
Population: All participants who received at least one dose of study drug who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Cohort 1: 100 mg LY2940680 | Cohort 2: 200 mg LY2940680 | Cohort 3: 400 mg LY2940680
Number analyzed (Participants) | 3 | 3 | 13
microgram per milliliter (µg/mL)
  LY2940680:Cycle 1 Day 1 | 0.841 (8) | 1.81 (5) | 3.84 (29)
  LY2940680:Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 10
  LY2940680:Cycle 1 Day 15 | 1.41 (51) | 3.10 (21) | 9.08 (40)
  LSN3185556:Cycle 1 Day 1 | 0.925 (45) | 1.49 (8) | 3.02 (30)
  LSN3185556:Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 10
  LSN3185556:Cycle 1 Day 15 | 2.12 (84) | 4.10 (22) | 13.7 (50)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From 0 to 24 Hours (AUC[0-24]) of LY2940680 and a Major Metabolite of LSN3185556
Description: Pharmacokinetics (PK): Area Under the Concentration time Curve From 0 to 24 Hours (AUC[0-24]) of LY2940680 and a Major Metabolite of LSN3185556.
Time Frame: Cycle1 Day1: Predose, 0.5,1,2,4, 6, 8, 10-12 hours; Cycle 1 Day15: Predose, 0.5,1,2,4, 6, 8, 10-12 hours
Population: All participants who received at least one dose of study drug who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter(µg*h/mL)
Arm/Group | Cohort 1: 100 mg LY2940680 | Cohort 2: 200 mg LY2940680 | Cohort 3: 400 mg LY2940680
Number analyzed (Participants) | 3 | 3 | 13
microgram*hour per milliliter(µg*h/mL)
  LY2940680:Cycle 1 Day 1 | 7.96 (31) | 20.3 (22) | 43.1 (26)
  LY2940680:Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 10
  LY2940680:Cycle 1 Day 15 | 14.7 (78) | 42.9 (40) | 142 (61)
  LSN3185556:Cycle 1 Day 1 | 13.2 (48) | 24.6 (5) | 50.1 (30)
  LSN3185556:Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 10
  LSN3185556:Cycle 1 Day 15 | 31.8 (126) | 79.7 (15) | 235 (48)

4. Secondary Outcome: Number of Participants Achieving Complete Response (CR) or Partial Response (PR) (Overall Response Rate[ORR])
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) criteria. CR was defined as the disappearance of all target and non-target lesions and all target and non-target lymph nodes were non-pathological or normal in size (<10 millimeter [mm] short axis). PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions taking as reference the baseline sum diameters. ORR calculated as: (sum of the number of participants with PRs and CRs) divided by (number of evaluable participants) multiplied by 100.
Time Frame: Baseline Until Disease Progression or Death Due to Any Cause (Up to 29 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 100 mg LY2940680 | Cohort 2: 200 mg LY2940680 | Cohort 3: 400 mg LY2940680
Number analyzed (Participants) | 3 | 3 | 13
Participants | 0 | 1 | 0

5. Secondary Outcome: Pharmacodynamic (PD): Percentage Change From Baseline in Gene Expression Level of Hedgehog (Hh) Regulated Genes (Gli1) in Skin
Description: Percentage Change From Baseline in Gene Expression Level of Hedgehog (Hh) Regulated Genes (Gli1) in Skin.
Time Frame: Baseline, Cycle 1 Day15
Population: All participants who received at least one dose of study drug and evaluable PD data.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort 1: 100 mg LY2940680 | Cohort 2: 200 mg LY2940680 | Cohort 3: 400 mg LY2940680
Number analyzed (Participants) | 3 | 2 | 10
percentage change | 92.73 (0.928) | 89.24 (2.096) | 92.86 (8.053)

ADVERSE EVENTS:
Time Frame: Baseline to End of Study (Up To 2.45 Years)
Arm/Group | Cohort 1: 100 mg LY2940680 | Cohort 2: 200 mg LY2940680 | Cohort 3: 400 mg LY2940680
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 4/13
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 100 mg LY2940680 (N=3) | Cohort 2: 200 mg LY2940680 (N=3) | Cohort 3: 400 mg LY2940680 (N=13)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 100 mg LY2940680 (N=3) | Cohort 2: 200 mg LY2940680 (N=3) | Cohort 3: 400 mg LY2940680 (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 9 (12)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 7 (8)
Fatigue (General disorders) | 1 (1) | 0 (0) | 10 (10)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (4)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram t wave inversion (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Mean cell haemoglobin concentration decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 10 (12)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2) | 8 (8)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days